CLINICAL TRIAL: NCT03489915
Title: Correlation Between the Visual Acuity and the OCT Pattern of Macular Edema Secondary to Retinal Vein Occlusion
Brief Title: Correlation Between the Visual Acuity & the OCT Pattern of Macular Edema Secondary to RVO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Omar Mohamed Ali, Resident, Assiut University
Other Study IDs: cbtvaatoctpomestrvo
Record Dates: First submitted 2018-03-23; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with macular edema due to RVO: assessment of visual acuity using Landolt chart and follow up of macular edema using OCT
  Interventions: Device: OCT

INTERVENTIONS:
Device: OCT — Assessment of macular edema secondary to retinal vein occlusion usin optical coherence tomography and its correlation with visual acuity

SUMMARY:
Correlation between changes observed in OCT and VA in patients with retinal vein occlusion whether the patient's VA improves when macular edema improves in OCT or not ??

DETAILED DESCRIPTION:
Central retinal vein occlusion (CRVO) is a common retinal vascular disorder. Clinically, CRVO presents with variable visual loss; fundus may show retinal hemorrhages, dilated tortuous retinal veins, cotton-wool spots, macular edIn view of the devastating complications associated with the severe form of CRVO, number of classifications were described. All of classifications take into account the area of retinal capillary nonperfusion and development of neovascular complications.

CRVO can be divided into 2 clinical types, ischemic and nonischemic. In addition, a number of patients may have an intermediate presentation with variable clinical course. On initial presentation, it may be difficult to classify a given patient, since CRVO may change with time.

A number of clinical and ancillary investigative factors are taken into account for classifying CRVO:

Nonischemic CRVO is milder form of disease. It may present with good vision, few retinal hemorrhages and cotton-wool spots, no relative afferent pupillary defect, and good perfusion to the retina. Nonischemic CRVO may resolve fully with good visual outcome or may progress to the ischemic type.

Ischemic CRVO is the severe form of the disease. CRVO may present initially as the ischemic type, or it may progress from nonischemic. Usually, ischemic CRVO presents with severe visual loss, extensive retinal hemorrhages and cotton-wool spots, presence of relative afferent pupillary defect, poor perfusion to retina, and presence of severe electroretinographic changes. In addition, patients may end up with neovascular glaucoma and a painful blind eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients with macular edema related to vein occlusion .
* Patient's Age above 18 years old .
* Patients able to sit on OCT device .

Exclusion Criteria:

* Significant cataract .
* Media opacities as vitreous haemorrhage .
* patients with macular edema related to CRVO treated by laser photocoagulation .
* patients with glaucoma .
* Patients with chronic uveitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in patients developing retinal vein occlusion for following up their changes in OCT & VA
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Macular edema assessment | 5 minutes
  Macular edema assessed by OCT in microns
Visual acuity assessment | 5 minutes
  Visual acuity assessment through Landolt chart

SECONDARY OUTCOMES:
Causes of non improvement of visual acuity in patients with resolving macular edema | 5 minutes
  To detect causes of visual non improvement with visual acuity measured through Landolt chart in patients with resolving macular edema measured by OCT device in microns

CONTACTS AND LOCATIONS:
Overall Officials: Abdelsalam a Mohamed, ass. prof., Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Natural history and clinical management of central retinal vein occlusion. The Central Vein Occlusion Study Group. Arch Ophthalmol. 1997 Apr;115(4):486-91. doi: 10.1001/archopht.1997.01100150488006. PMID 9109757
- [Background] Hayreh SS. Classification of central retinal vein occlusion. Ophthalmology. 1983 May;90(5):458-74. doi: 10.1016/s0161-6420(83)34530-9. PMID 6877778
- [Background] Hayreh SS. Retinal vein occlusion. Indian J Ophthalmol. 1994 Sep;42(3):109-32. PMID 7829175
- [Background] Williamson TH. Central retinal vein occlusion: what's the story? Br J Ophthalmol. 1997 Aug;81(8):698-704. doi: 10.1136/bjo.81.8.698. No abstract available. PMID 9349161
- [Result] Hayreh SS, Zimmerman MB, Podhajsky P. Incidence of various types of retinal vein occlusion and their recurrence and demographic characteristics. Am J Ophthalmol. 1994 Apr 15;117(4):429-41. doi: 10.1016/s0002-9394(14)70001-7. PMID 8154523
- [Result] Moschos MM, Moschos M. Intraocular bevacizumab for macular edema due to CRVO. A multifocal-ERG and OCT study. Doc Ophthalmol. 2008 Mar;116(2):147-52. doi: 10.1007/s10633-007-9110-9. Epub 2008 Jan 10. PMID 18189152
- [Result] Gupta B, Grewal J, Adewoyin T, Pelosini L, Williamson TH. Diurnal variation of macular oedema in CRVO: prospective study. Graefes Arch Clin Exp Ophthalmol. 2009 May;247(5):593-6. doi: 10.1007/s00417-008-1011-4. Epub 2008 Dec 4. PMID 19052771